CLINICAL TRIAL: NCT00666783
Title: A Phase II, Multicenter,Double-Blind, Randomized Trial of Palonosetron Compared With Granisetron in Preventing Highly Emetogenic Chemotherapy-Induced Nausea and Vomiting in the Chinese Cancer Patients
Brief Title: An Efficacy and Safety Study of Palonosetron in Preventing Chemotherapy-Induced Nausea and Vomiting (CINV) in the Chinese Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Xijing Hospital, Clinical trial center of Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2006L01595
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2006-08

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Palonosetron; Granisetron

ARMS (2):
- PAL (Experimental): receive any of the following cytotoxic agents based combination chemotherapy (epirubicin 60 mg/m2, or cisplatin 75 mg/m2)
  Interventions: Drug: palonosetron
- GRA (Active Comparator): receive any of the following cytotoxic agents based combination chemotherapy (epirubicin 60 mg/m2, or cisplatin 75 mg/m2)
  Interventions: Drug: Granisetron

INTERVENTIONS:
Drug: palonosetron — receive a single, intravenous dose of palonosetron 0.25 mg, 30 minutes before receiving highly emetogenic chemotherapy.
  Arms: PAL
Drug: Granisetron — receive a single, intravenous dose of granisetron 3 mg, 30 minutes before chemotherapy.
  Arms: GRA

SUMMARY:
This clinical study was designed to demonstrate that a single, intravenous dose of palonosetron 0.25 mg was not inferior to granisetron 3 mg in preventing acute and delayed CINV and was also well tolerated in the Chinese cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ranging from 18 yrs to 70 yrs, with histologically or cytologically confirmed malignant disease
* naive to chemotherapy or nonnaive with an interval of at least 14 days to the last one
* Karnofsky index more than 70% and anticipated survival time more than 90 days
* Scheduled to receive any of the following cytotoxic agents based combination chemotherapy (epirubicin 60 mg/m2, or cisplatin 75 mg/m2) on study Day 1 and the chemotherapy should be accomplished on study Day 1
* No emetic episodes and antiemetic medication during the 24 hours preceding chemotherapy administration
* Adequate organ functions(No impairment to renal, hepatic, cardiac or bone marrow function )
* Use of reliable contraceptive measures (for females of childbearing potential) and negative pregnancy test at baseline visit
* Provision of written informed consent

Exclusion Criteria:

* Inability to understand or cooperate with study procedures
* Receipt of investigational drugs 30 days before study entry
* Scheduled to receive any drug with antiemetic efficacy from 24 hrs before to 5 days after treatment
* Contraindications to 5-HT3 receptor antagonists
* Woman Patient with Pregnancy or lactation
* Diagnosed with hypertension or severe infectious diseases
* Obstructive symptom of gastrointestinal tract
* Symptomatic brain metastasis or mental dysfunction
* Baseline QTc > 500 ms

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Xijng Hospital, Xi'an, Shaanxi, China